CLINICAL TRIAL: NCT04019002
Title: Evaluating Hyperpolarized and Proton Brain Metabolism in Patients With Glioblastoma
Brief Title: Hyperpolarized Carbon-13 (13C) Pyruvate Imaging in Patients With Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Susan Chang (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Susan Chang, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19105; 2P50CA097257 (NIH); NCI-2019-07406 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: Glioblastoma Multiforme; Hyperpolarized Pyruvate; Magnetic Resonance; Magnetic Resonance Spectroscopic Imaging; Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Newly Diagnosed- Standard Treatment (Experimental): This arm is for patients with histologically proven newly diagnosed glioblastoma who will undergo standard treatment with radiation therapy (RT) and temozolomide (TMZ).
  Patients will receive two injections of hyperpolarized 13C pyruvate for research imaging performed prior to standard imaging on the same day. Research imaging occurs at two time points: before receiving standard treatment with RT/TMZ and at the first post-radiation follow-up scan (8 weeks later).
  Interventions: Drug: Hyperpolarized 13C Pyruvate
- Cohort 2: Recurrent- Standard Surgical Resection (Experimental): This arm is for patients with histologically proven recurrent suspected glioblastoma who will receive surgical resection for the recurrence.
  Patients will receive one injection of hyperpolarized 13C pyruvate for research imaging performed prior to standard imaging on the same day. Research imaging occurs at one time point: before surgery.
  Interventions: Drug: Hyperpolarized 13C Pyruvate
- Cohort 3: Recurrent- Standard Treatment (Experimental): This arm is for patients with histologically proven recurrent suspected glioblastoma who will undergo standard treatment for the recurrence.
  Patients will receive two injections of hyperpolarized 13C pyruvate for research imaging performed prior to standard imaging on the same day. Research imaging occurs at three time points: prior to treatment (baseline), approximately 7-14 days after the initiation of treatment, and 6-8 weeks after the initiation of treatment.
  Interventions: Drug: Hyperpolarized 13C Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C Pyruvate — Given at 0.43 milliliters/kilogram body weight of a 250 millimolar (mM) solution via intravenous injection over a period of about 1 minute once prior to each research magnetic resonance imaging procedure.
  Other Names: HP-13C

SUMMARY:
The purpose of this study is to evaluate whether new metabolic imaging will be useful to physicians and patients with glioblastoma for making treatment decisions and seeing how well various types of treatment work. The goal is to improve the way patient care is managed in the future.

If you chose to be in this study, you will be receiving novel magnetic resonance (MR) metabolic imaging with standard MR imaging. The research component includes an injection of an investigational agent, called hyperpolarized 13C pyruvate, to obtain dynamic metabolic imaging.

DETAILED DESCRIPTION:
The new metabolic imaging will use hyperpolarized 13C pyruvate, which allows for pictures of the brain that we won't be able to get with standard imaging. Hyperpolarized 13C pyruvate has not been approved for use by the Food and Drug Administration (FDA) and is available for research only. This investigational agent is a non-radioactive isotope of carbon.

There are three groups in this study. Assignment to a study group depends on the status of your disease and the type of treatment you will be receiving.

Subjects in Group 1 will have two MR examination time points. Each time point includes a hyperpolarized 13C pyruvate injection for research imaging as well as standard MR. The MR examinations will occur before receiving standard of care treatment with radiation and chemotherapy, and at the first post-radiation follow-up scan.

Subjects in Group 2 will have one MR examination time point with hyperpolarized 13C pyruvate injection for research and standard MR. This MR examination occurs before surgery.

Subjects in Group 3 will have three MR examination time points. Each time point includes a hyperpolarized 13C pyruvate injection for research imaging as well as standard MR. The MR examinations will occur prior to initiating therapy (baseline), at approximately 7-14 days after initiation of therapy, and 6-8 weeks after the initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Histologically proven newly diagnosed glioblastoma multiforme (GBM) who will undergo standard of treatment with radiation therapy (RT) and temozolomide (TMZ).
* Cohort 2: Histologically proven recurrent suspected GBM who will receive surgical resection for the recurrence.
* Cohort 3: Histologically proven recurrent suspected GBM who will undergo standard treatment for the recurrence.
* Patients must be >/= 18 years old and with a life expectancy > 16 weeks.
* Patients must have a Karnofsky performance status of ≥ 70.
* Patients must have adequate renal function: creatinine < 1.5 mg/dL before imaging. These tests must be performed within 60 days prior to Hyperpolarized Imaging scan.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to tolerate the imaging examination or any disease that will obscure toxicity or dangerously alter response to the imaging agent.
* Patients must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Patients must not have a history of myocardial infarction or unstable angina within 12 months prior to study enrollment.
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. Minorities will actively be recruited to participate. No exclusion to this study will be based on race.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must sign an authorization for the release of their protected health information.
* Patients may not be known to be human immunodeficiency virus (HIV)-positive. HIV testing is not required for study participation.
* Patients must not have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* Patients must not be pregnant or breast feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of Hyperpolarized Imaging scan. Effective contraception (men and women) must be used in subjects of child-bearing potential.

Exclusion Criteria:

* Subjects must be excluded from participating in this study if they are not able to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (AEs) Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | From Day 1 through study completion, up to 4 months
  Patients will be monitored for the occurrence of AEs that occur during the course of study participation. AE monitoring occurs on each day of hyperpolarized 13C pyruvate administration and until 7 days after administration. Serious adverse events occurring more than 7 days after administration need only be reported if relationship to the investigational drug is suspected.
Number of Dose-Limiting Toxicities (DLTs) Assessed by CTCAE Version 4.0 | From Day 1 through study completion, up to 4 months
  A DLT for this protocol is defined as any event grade 3 or higher in severity assessed by CTCAE version 4.0 that is possibly, probably, or definitely attributable to the investigational drug, excluding laboratory abnormalities determined to be clinically insignificant.
Describe Changes in 13C pyruvate-to-lactate conversion rate (kPL) in Normal and Diseased Brain Tissues | Day 1 and Week 8
  The changes in 13C kPL from baseline to the post-RT scan will be compared in the normal appearing brain, enhancing lesion, and non-enhancing lesion
Describe Changes in 13C Lactate/Pyruvate Ratio in Normal and Diseased Brain Tissues | Day 1 and Week 8
  The changes in 13C lactate/pyruvate ratio from baseline to the post-RT scan will be compared in the normal appearing brain, enhancing lesion, and non-enhancing lesion
Compare 13C kPL Between Recurrent Lesions and Regions of Treatment Related Effects | Day 1, Week 1-2, and Week 6-8
  The 13C kPL from the recurrent lesions will be compared to those in the regions of treatment related effects.
Compare 13C Lactate/Pyruvate Ratio Between Recurrent Lesions and Regions of Treatment Related Effects | Day 1, Week 1-2, and Week 6-8
  The 13C lactate/pyruvate ratio from the recurrent lesions will be compared to those in the regions of treatment related effects.
Determine the Association Between 13C kPL and Time to Disease Progression | From Day 1 until the date of documented disease progression, an average of 1 year
  Relationships between 13C kPL and time to disease progression will be compared. Time to disease progression is defined as the time from first study imaging until worsening of glioblastoma disease.
Determine the Association Between 13C Lactate/Pyruvate Ratio and Time to Disease Progression | From Day 1 until the date of documented disease progression, an average of 1 year
  Relationships between 13C lactate/pyruvate ratio and time to disease progression will be compared. Time to disease progression is defined as the time from first study imaging until worsening of glioblastoma disease.
Determine the Association Between Hydrogen-1 (1H) Choline-to-N-acetylaspartate (NAA) index (CNI) and Time to Disease Progression | From Day 1 until the date of documented disease progression, an average of 1 year
  Relationships between 1H CNI time to disease progression will be compared. Time to disease progression is defined as the time from first study imaging until worsening of glioblastoma disease.
Determine the Association Between 13C kPL and Overall Survival | From Day 1 until the date of death from any cause, up to 2 years
  Relationships between 13C kPL and overall survival will be compared. Overall Survival is defined as the time from first study imaging until death from any cause.
Determine the Association Between 13C Lactate/Pyruvate Ratio and Overall Survival | From Day 1 until the date of death from any cause, up to 2 years
  Relationships between 13C lactate/pyruvate ratio and overall survival will be compared. Overall Survival is defined as the time from first study imaging until death from any cause.
Determine the Association Between 1H CNI and Overall Survival | From Day 1 until the date of death from any cause, up to 2 years
  Relationships between 1H CNI and overall survival will be compared. Overall Survival is defined as the time from first study imaging until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04019002/ICF_000.pdf